CLINICAL TRIAL: NCT07164027
Title: Beacon: Prospective Assessment of Flotufolastat F 18 PSMA and MRI in the Diagnosis of Clinically Significant Prostate Cancer
Brief Title: Comparing a New PSMA Imaging Agent to MRI for Detecting Prostate Cancer, BEACON Trial
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-1372; NCI-2025-05056 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Masking Description: Nuclear medicine physicians will initially be blinded to MRI findings while interpreting and outlining the PSMA PET/CT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (flotufolastat F-18 PET/CT) (Experimental): Patients receive flotufolastat F-18 IV and then, 50-100 minutes later, undergo PET/CT over 30 minutes. Within 6 months of PET/CT imaging, patients undergo PSMA PET/CT/US fusion biopsy and MRI/US fusion biopsy in a randomized order. Patients may undergo blood sample collection at screening and/or on study.
  Interventions: Procedure: Biopsy of Prostate; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Flotufolastat F-18 Gallium; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Radiation: Flotufolastat F-18 Gallium — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 Radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; Posluma; rhPSMA-7.3 (18F)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This early phase I trial evaluates whether a new imaging technique using flotufolastat F 18 (a type of prostate specific membrane antigen [PSMA] imaging agent) with positron emission tomography (PET)/computed tomography (CT) can be used to guide targeted prostate biopsies in men with prostate cancer. Flotufolastat F 18 is a radioactive imaging agent that binds to prostate tumor cells that express PSMA. This allows for visualization of PSMA-expressing tumor cells on imaging scans such as PET/CT. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, flotufolastat F 18. Because prostate cancer takes up flotufolastat F 18, it can be seen with PET. CT utilizes X-rays that track the body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in the body. The PET/CT scanner combines the PET and the CT scanners into a single device. A targeted prostate biopsy refers to using advanced imaging for guidance when taking samples (biopsies) of the prostate. This method can fuse (combine) PET/CT images with real-time ultrasound during a prostate biopsy. PSMA PET/CT scans have the potential for guiding prostate biopsies. Using image fusion technology, they can increase detection of prostate cancer by providing anatomical information and guidance during a prostate biopsy. Improved detection of prostate cancer using PSMA PET/CT guidance may better inform men and their clinicians about prostate cancer risk and management. This study attempts to determine how often prostate cancer is found when using PSMA PET/CT scan images during a biopsy versus the conventional magnetic resonance imaging-guidance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the detection rate of flotufolastat F 18 and magnetic resonance imaging (MRI) regions of interest for grade group 2 and greater prostate cancer.

SECONDARY OBJECTIVES:

I. Evaluate the detection rate of incidental grade group (GG)1 prostate cancer (region of interest [ROI] benign, systematic GG1).

II. Evaluate the patient-level GG ≥ 2 detection rate for increasing standardized uptake value (SUV) and Prostate Imaging-Reporting and Data System (PI-RADS) score to determine if/when systematic biopsy may be omitted.

III. Evaluate the concordance between biopsy methods for intraprostatic tumor location (e.g., right versus [vs.] left vs. bilateral).

IV. Validate the MRI + prostate specific membrane antigen (PSMA)-positron emission tomography (PET) composite (P) score for prostate biopsy.

EXPLORATORY OBJECTIVES:

1. Evaluate if MRI vs PSMA ROI detects more aggressive cancer clones based on the percentage of Gleason pattern 4 or 5.
2. Compare the tumor volume of PSMA and MRI for men proceeding to focal therapy.

OUTLINE:

Patients receive flotufolastat F-18 intravenously (IV) and then, 50-100 minutes later, undergo PET/CT over 30 minutes. Within 6 months of PET/CT imaging, patients undergo PSMA PET/CT/ultrasound (US) fusion biopsy and MRI/US fusion biopsy in a randomized order. Patients may undergo blood sample collection at screening and/or on study.

After completion of study intervention, patients are followed up within 3 months of their biopsy and then every 12 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-90 at study enrollment
* Have at least one PI-RADS 3-5 lesion on MRI within the 12 months prior to enrollment

Exclusion Criteria:

* Contraindication to flotufolastat F 18 PET CT
* Contraindication to ultrasound-guided prostate biopsy
* Previous treatment of prostate cancer
* Unable to discontinue blood thinners for 7 days prior to biopsy
* Any investigational agents within 42 days prior to the day of the first dose
* Not able to understand and to follow study instructions and requirements. This also includes the inability to complete the study imaging and or biopsy procedures due to any reason (e.g., severe claustrophobia, inability to lie still for the entire imaging time, any condition that precludes raised arms position)

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2036-01-28 (Estimated); Study Completion 2037-01-28 (Estimated)

PRIMARY OUTCOMES:
Detection of high-grade cancer (grade group [GG] ≥ 2) | At time of biopsy
  Results of prostate specific membrane antigen (PSMA)- and magnetic resonance imaging (MRI)-guided biopsy will be compared to the results of systematic biopsy in the same patient.

SECONDARY OUTCOMES:
Proportion of subjects with incidental GG1 prostate cancer detected through systematic biopsy when the region of interest is benign on MRI and PSMA-positron emission tomography (PET) | At time of biopsy
Rate of detection of GG ≥ 2 prostate cancer in relation to increasing standardized uptake value and Prostate Imaging-Reporting and Data System scores | At time of biopsy
Percentage of cases where the intraprostatic tumor location identified by MRI-guided and PSMA-guided biopsies matches | At time of biopsy
Accuracy and predictive value of the MRI + PSMA-PET composite score for detecting clinically significant prostate cancer during biopsy | At time of biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Brisbane, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States